CLINICAL TRIAL: NCT06921993
Title: Lung Ultrasound for Antibiotic Stewardship in Community-Acquired Pneumonia: A Randomized Clinical Trial
Brief Title: Lung Ultrasound for Guiding Antibiotic Use in Pediatric Pneumonia
Acronym: LUSCAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Gaslini Children's Hospital (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); University Hospital Padova (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other); Bambino Gesù Hospital and Research Institute (Other); Santobono-Pausilpon Hospital (Unknown); Asst Degli Spedali Civili Di Brescia (Other); IRCCS Burlo Garofolo (Other); Clinica Pediatrica Università di Novara (Unknown); Hospital of Prato (Other); Columbia University (Other); Schneider Children's Medical Center, Israel (Other); Yale University (Other); University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LUSCAP
Record Dates: First submitted 2025-04-02; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pneumonia Childhood; Pneumonia; Lung Ultrasound; Antibiotic Stewardship
Keywords: Pneumonia; Children; Pediatrics; Lung ultrasound; point-of-care ultrasound
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: Randomized diagnostic clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group - standard of care (No Intervention): All subjects randomly assigned to the control arm will undergo a complete patient history and clinical assessment (the reference standard). If there is clinical uncertainty, the enrolling physician has the option to perform other test such as CXR or blood test.
- Experimental Group - Lung Ultrasound (LUS) (Experimental): All subjects randomly assigned to the investigational arm will undergo lung ultrasound (LUS) . The LUS will be performed immediately following a thorough patient history and complete clinical assessment.
  Ultrasound still images and ultrasound clips will be acquired according to the study protocol. Detailed methodology of the ultrasound examination and parameters is provided as appendix to the study protocol
  Interventions: Diagnostic Test: LUNG ULTRASOUND

INTERVENTIONS:
Diagnostic Test: LUNG ULTRASOUND — All subjects randomly assigned to the investigational arm will undergo lung ultrasound (LUS) .
  Ultrasound still images and ultrasound clips will be acquired according to the study protocol. Detailed methodology of the ultrasound examination and parameters is provided as appendix to the study protocol
  Arms: Experimental Group - Lung Ultrasound (LUS)

SUMMARY:
Pneumonia is a major cause of illness and death in children, with an annual incidence of about 3.3 per 1,000 in those under five years old, many requiring hospitalization. The diagnosis is challenging due to the absence of a universally accepted gold standard, leading to variability in emergency settings. Current guidelines recommend diagnosis based on history and physical examination, which do not reliably differentiate pneumonia from other respiratory infections or identify whether it is bacterial or viral in nature. This uncertainty can lead to the unnecessary use of antibiotics.

Commonly used chest X-rays have limitations such as low sensitivity, moderate interobserver reliability, and the inability to distinguish bacterial from viral pneumonia. In contrast, lung ultrasound has shown high sensitivity and specificity for diagnosing pneumonia in children. However, lung ultrasound also cannot reliably distinguish between bacterial and viral causes and might lead to increased antibiotic prescriptions by detecting minor lung consolidations not seen on chest X-rays. Despite these issues, lung ultrasound is widely used in pediatric pulmonary assessment.

The primary objective of the study is to determine if using lung ultrasound for diagnosing pneumonia in children can reduce antibiotic prescriptions compared to the standard care approach-which mainly relies on clinical diagnosis (often supplemented by chest X-ray and blood tests in selected cases). The secondary objective is to assess how frequently lung ultrasound impacts management decisions during a single clinical visit, beyond the information provided by history and physical examination. The third objective is to compare the diagnostic accuracy of lung ultrasound-supported diagnosis with existing diagnostic methods.

The study hypothesizes that lung ultrasound results can act as a decision modifier, similar to other clinical tools and examination findings. However, a lack of consensus on specific lung ultrasound parameters and their clinical correlations contributes to variability in managing suspected pneumonia, potentially leading to antibiotic overuse.

Eligible participants are children aged three to ten years who are in good general condition and clinically stable, presenting with signs and symptoms of lower respiratory tract infection indicative of pneumonia. Exclusion criteria include children outside the specified age range, those recently hospitalized, those who have undergone prior chest imaging, those already on antibiotic therapy, those with severe clinical instability, and those with underlying conditions predisposing them to severe or recurrent pneumonia. These criteria help ensure that the study population represents general pediatric community-acquired pneumonia cases, avoiding biases from high-risk patients.

The ultimate goal of this study is to provide evidence on whether lung ultrasound can serve as a reliable tool to guide antibiotic prescriptions, thereby reducing unnecessary antibiotic use in the management of pediatric pneumonia.

DETAILED DESCRIPTION:
This prospective, randomized, multicenter clinical trial aims to determine whether using lung ultrasound (LUS) in children aged 3-10 years with suspected pneumonia can reduce the prescription of antibiotics, compared to the standard of care (clinical diagnosis, with optional chest X-ray and blood tests). A second objective is to assess how often LUS findings alter clinical decision-making beyond history and physical examination alone, while a third objective compares the diagnostic accuracy of an LUS-based approach to current pathways.

Study Design and Intervention

Children presenting with signs and symptoms of lower respiratory tract infection (e.g., cough, tachypnea, fever) who are clinically stable and in good general condition are eligible.

Exclusion criteria include recent hospitalization, prior imaging, ongoing antibiotic therapy, severe respiratory distress, and underlying conditions predisposing to complicated pneumonia.

Participants are randomized to an experimental group, where LUS is performed immediately after clinical assessment, or a control group, which follows standard care.

Clinicians in both groups may request a chest X-ray if warranted, and the reasons for imaging are documented.

All participants receive routine evaluations, and interventions (e.g., blood tests, antibiotic decisions) remain at the discretion of the treating physician.

Outcomes

Primary Outcome: Reduction in antibiotic prescriptions in the LUS group versus the control group.

Secondary Outcomes:

The rate at which LUS modifies diagnoses and clinical management compared to assessments using only history and physical examination.

Differences in emergency department (ED) length of stay, hospital admission rates, and unscheduled healthcare visits within one week.

Overall diagnostic accuracy of LUS-supported diagnosis compared to standard methods.

Additional Measures:

An expert panel (pediatric radiologist, pulmonologist, and emergency physician) will determine a consensus final diagnosis after reviewing clinical data.

Data Management and Follow-Up

Each patient's care pathway is documented using a 1-5 Likert scale capturing the likelihood of pneumonia and willingness to prescribe antibiotics at various decision points (clinical exam, optional LUS, and optional chest X-ray).

A follow-up call occurs 5-7 days post-discharge to track clinical progress and any subsequent antibiotic use.

Data are recorded and stored in REDCap, with pseudonymized patient identifiers.

No significant risks are anticipated. The benefits include potentially improving diagnostic accuracy and reducing unnecessary antibiotic prescriptions.

Ultimately, this study seeks to clarify whether incorporating LUS into standard pediatric pneumonia assessment can enhance decision-making, leading to more judicious antibiotic use without compromising patient care.

ELIGIBILITY:
Inclusion Criteria:

* Well-appearing, clinically stable patients aged 3 to 10 years, presenting to the pediatric ED with suspected pneumonia based on a combination of signs and symptoms suggestive of lower respiratory tract infection (LRTI), including:

  1. Respiratory Symptoms: Cough, Tachypnea, Dyspnea (Increased work of breathing), Abnormal findings on auscultation.
  2. Systemic Symptoms: Fever, Hypoxia, Decreased appetite.

     Exclusion Criteria:
* Neonates and children up to 3 years of age, and children older than 10 years
* Children aged 3 to 10 years with any of the following factors:

  1. Recent hospitalization (within the past 14 days)
  2. Prior CXR or any other chest imaging (e.g. CT scan)
  3. Ongoing antibiotic therapy
  4. Hemodynamic instability
  5. Respiratory failure or severe respiratory distress and/or hypoxemia, requiring urgent assessment for conditions such as pneumothorax, hemothorax, or other emergency respiratory conditions
  6. History of aspiration or ab ingestis pneumonia
  7. Underlying medical conditions predisposing to severe or recurrent pneumonia, including immunodeficiency, chronic corticosteroid use, chronic lung disease, malignancy, sickle cell disease, congenital heart disease, tracheostomy, and neuromuscular disorders affecting respiration

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 659 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with antibiotic use | 7 days
  A chart review and follow up phone call made at 1 week (range 5-7 days) to assess whether or not the subject was started on antibiotics during the index ED visit or at a later healthcare visit. The primary objective of this study is to determine if it is possible for LUS to reduce antibiotic prescription when evaluating patients with possible pneumonia. Specifically, an overall reduction of antibiotic when LUS is used as adjunct tool in the

SECONDARY OUTCOMES:
Percentage of participants who had hospital admission | 7 days
  Chart review and follow up phone call made at 1 week (range 5-7 days) to assess whether or not the subject was admitted during the index ED visit or at a later healthcare visit.
Percentage of participants with antibiotic use | 7 days
  A chart review and follow up phone call made at 1 week (range 5-7 days) to assess whether or not the subject was started on antibiotics during the index ED visit or at a later healthcare visit. The primary objective of this study is to determine if it is possible for LUS to reduce antibiotic prescription when evaluating patients with possible pneumonia. Specifically, an overall reduction of antibiotic when LUS is used as adjunct tool in the assessment.

OTHER OUTCOMES:
Percentage of Participants Whose Pneumonia Was Missed by LUS or CXR | 30 days
  Diagnostic accuracy of the 2 different imaging techniques
Comparison of Unscheduled Healthcare Visits | 7 days
  Percentage of participants who had unscheduled healthcare visits after the index ED visit between those subjects who undergo CXR first and those who undergo LUS first.
Comparison of the Length of Stay in the emergency department | day 1
  Chart review conducted to assess overall length of stay in the ED.

CONTACTS AND LOCATIONS:
Overall Officials: Niccolò Parri, MD, Study Director — Meyer Children's Hospital IRCCS, Florence, Italy
Locations (1):
- Meyer Children's Hospital IRCCS, Florence, Italy, Italy

IPD SHARING:
Plan to Share IPD: No